CLINICAL TRIAL: NCT03878446
Title: A Dose-finding Trial Evaluating the Effect and Safety of Once-weekly Treatment of Somapacitan Compared to Daily Norditropin® in Children With Short Stature Born Small for Gestational Age With no Catch-up Growth by 2 Years of Age or Older
Brief Title: A Research Study in Children Born Small and Who Stayed Small. Treatment is Somapacitan Once a Week Compared to Norditropin® Once a Day
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NN8640-4245; U1111-1207-9741 (Other: World Health Organization (WHO)); 2018-000232-10 (EudraCT Number)
Record Dates: First submitted 2019-03-15; First posted 2019-03-18 (Actual); Results first posted 2024-06-20 (Actual); Last update posted 2025-12-23 (Actual); Status verified 2025-12

CONDITIONS: Short Stature Children Born Small for Gestational Age (SGA)
MeSH Terms: interventions — somapacitan; Human Growth Hormone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- Somapacitan 0.24 mg/kg/week (Experimental): Same treatment in main period (26 weeks) and extension period I (26 weeks). Dosage of Somapacitan during extension period II will be determined based on the data from main phase.
  Interventions: Drug: Somapacitan
- Somapacitan 0.20 mg/kg/week (Experimental): Same treatment in main period (26 weeks) and extension period I (26 weeks). Dosage of Somapacitan during extension period II will be determined based on the data from main phase.
  Interventions: Drug: Somapacitan
- Somapacitan 0.16 mg/kg/week (Experimental): Same treatment in main period (26 weeks) and extension period I (26 weeks). Dosage of Somapacitan during extension period II will be determined based on the data from main phase.
  Interventions: Drug: Somapacitan
- Norditropin® 0.035 mg/kg/day (Active Comparator): Same treatment in main period (26 weeks) and extension period I (26 weeks). Participants will switch to Somapacitan during extension period II. Dosage of Somapacitan during extension period II will be determined based on the data from main phase.
  Interventions: Drug: Norditropin®
- Norditropin® 0.067 mg/kg/day (Active Comparator): Same treatment in main period (26 weeks) and extension period I (26 weeks). Participants will switch to Somapacitan during extension period II. Dosage of Somapacitan during extension period II will be determined based on the data from main phase.
  Interventions: Drug: Norditropin®

INTERVENTIONS:
Drug: Somapacitan — Somapacitan injected under the skin once a week.
  Arms: Somapacitan 0.16 mg/kg/week; Somapacitan 0.20 mg/kg/week; Somapacitan 0.24 mg/kg/week
Drug: Norditropin® — Norditropin® injected under the skin once a day.
  Arms: Norditropin® 0.035 mg/kg/day; Norditropin® 0.067 mg/kg/day

SUMMARY:
The study compares 2 medicines used for the treatment of children who are born small and who stayed small: somapacitan given once a week (a new medicine) and Norditropin® given once a day (the medicine doctors can already prescribe).

Participants will either get somapacitan or Norditropin® - which treatment is decided by chance. Both participants and the study doctor will know which treatment the participants get. The study will last for 5 years. Participants will take either an injection once every week or once every day.

ELIGIBILITY:
Inclusion Criteria:

* Pre-pubertal children, boys:

  1. age between 2.5 and 11.0 years at screening.
  2. testes volume below 4 ml.
* Pre-pubertal children, girls:

  1. age between 2.5 and 10.0 years at screening.
  2. Tanner stage 1 for breast development (no palpable glandular breast tissue).
* Born small for gestational age (birth length and/or weight below -2 standard deviation scores) (according to national standards).
* Impaired height defined as at least 2.5 standard deviations below the mean height for chronological age and gender at screening according to the standards of Centers for Disease Control and Prevention at screening.
* Impaired height velocity defined as annualized height velocity below the 50th percentile for chronological age and gender according to the standards of Prader calculated over a time span of minimum 6 months and maximum 18 months prior to screening.
* No prior exposure to growth hormone therapy or Insulin-like Growth Factor-I (IGF-I) treatment.

Exclusion Criteria:

* Any known or suspected clinically significant abnormality likely to affect growth or the ability to evaluate growth with standing height measurements.
* Children with hormonal deficiencies including suspected or confirmed growth hormone deficiency according to local practise.
* Current inflammatory diseases requiring systemic corticosteroid treatment for longer than 2 consecutive weeks within the last 3 months prior to screening.
* Children requiring inhaled glucocorticoid therapy at a dose of greater than 400 μg/day of inhaled budesonide or equivalents for longer than 4 consecutive weeks within the last 12 months prior to screening.
* Concomitant administration of other treatments that may have an effect on growth, e.g but not limited to methylphenidate for treatment of attention deficit hyperactivity disorder.
* Diagnosis of attention deficit hyperactivity disorder.
* Prior history or presence of malignancy including intracranial tumours.

Ages: 2 Years to 11 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 62 (Actual)
Dates: Start 2019-07-04 (Actual); Primary Completion 2021-05-05 (Actual); Study Completion 2026-12-23 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Reporting Anchor and Disclosure 1452, Study Director — Novo Nordisk A/S
Locations (92):
- United States (14):
  - Univ of AL at Birmingham_BRM, Birmingham, Alabama
  - Children's Hosp Of Orange, Orange, California
  - St. Luke's Children's Endo, Boise, Idaho
  - Univ of Minnesota M.C.H., Minneapolis, Minnesota
  - Children's Minnesota, Saint Paul, Minnesota
  - Goryeb Children's Hospital, Morristown, New Jersey
  - Rutgers-Rwjms, New Brunswick, New Jersey
  - NYU Langone Hospital-LI, Garden City, New York
  - NYU Langone Hospital-LI, Mineola, New York
  - Icahn Sch of Med-Mt Sinai Hosp, New York, New York
  - CCHMC_Cinc, Cincinnati, Ohio
  - Univ Oklahoma Sci Ctr OK City, Oklahoma City, Oklahoma
  - Cook Children's Hospital-Hematology-Oncology, Fort Worth, Texas
  - MultiCare Inst for Res & Innov, Tacoma, Washington
- Algeria (3):
  - CHU Bab El Oued Pediatrics Dept, Algiers
  - Endo and Diab Dept El Oued, Algiers
  - endocrino-diabetology department, Hospital IBN BADIS., Constantine
- Austria (5):
  - Kepler Universitätsklinikum GmbH - Med Campus IV (vorm.LFKK), Linz, Upper Austria
  - Med. Univ. Graz -Klinische Abteilung f. Allgemeine Pädiatrie, Graz
  - LKH Salzburg- Univ. Klinik f. Kinder- und Jugendheilkunde, Salzburg
  - LKH St. Poelten, Kinder-und Jugendheilkunde, Sankt Pölten
  - Salzkammergut-Klinikum Vöcklabruck, Vöcklabruck
- Stollery Children's Hospital, Edmonton, Alberta, Canada
- Rigshospitalet Klinik for Vækst og Reproduktion Afsnit 5064, Copenhagen Ø, Denmark
- Estonia (2):
  - Tallinn Children's Hospital, Tallinn
  - Tartu University Hospital Children's Clinic, Tartu
- France (7):
  - Centre Hospitalier Universitaire D'Angers-2, Angers
  - Ap-Hp-Hopital de Bicetre-2, Le Kremlin-Bicêtre
  - Assistance Publique Hopitaux de Marseille-Hopital de La Timone-2, Marseille
  - Hopital de La Timone, Marseille Cédex 05
  - Ap-Hp-Hopital Necker-2, Paris
  - Hôpital Necker, Paris
  - Hopital Des Enfants-2, Toulouse
- Hungary (2):
  - Észak-Közép-budai Centrum, Szent János Kórház és Szakrendelő, Budapest
  - Szegedi Tudományegyetem Gyermekgyógyászati Klinika, Szeged
- India (3):
  - Amrita Institute Of Medical Sciences & Research Centre, Kochi, Kerala
  - Jehangir Clinical Development Centre, Pune, Maharashtra
  - All India Institute of Medical Sciences, New Dehli, New Delhi
- CHI Crumlin Dept of Endocrinology, Dublin, Ireland
- Israel (3):
  - Rambam MC - Department of Pediatrics A, Haifa
  - Meir MC - Department of Paediatrics, Kfar Saba
  - Schneider MC - Endrocrinology and Diabetes, Petah Tikva
- Italy (4):
  - IRCCS Meyer Firenze, Florence
  - Ospedale Pediatrico Gaslini, Genova
  - Ospedale Maggiore Policlinico UO Endocrinologia Diabetolgia, Milan
  - Ospedale Pediatrico Bambino Gesu, Roma
- Japan (15):
  - Kurume University Hospital, Pediatrics, Fukuoka
  - Fukuoka Children's Hospital_Endocrinology and Metabolism, Fukuoka-shi, Fukuoka
  - Fukuoka Children's Hospital, Fukuoka-shi, Fukuoka
  - Fukuyama City Hospital_Department of Pediatrics, Fukuyama-shi, Hiroshima
  - Hyogo Prefectual Kobe Children's Hospital Dept. Metab & endo, Kobe-shi, Hyogo
  - Univ.HP, Kyoto Pref Univ of Medicine, Dept. of Pediatrics, Kyoto
  - Nara Prefecture General Medical Center_ Nara-shi, Nara, Nara-shi, Nara
  - Niigata University Medical & Dental Hospital_Pediatrics, Niigata-shi, Niigata
  - Osaka City General Hospital, Pediatric Endocrinology and Me, Osaka
  - Osaka Women's and Children's Hospital, Osaka
  - Saitama Children's Medical Center, Endocrinorogy&Metabolism, Saitama-shi, Saitama
  - Institute of Science Tokyo Hospital_Pediatrics, Tokyo
  - Institute of Science Tokyo Hospital, Tokyo
  - National Center for Child Health and Dev, Endo and Metabo, Tokyo
  - Keio University Hospital, Pediatrics, Tokyo
- Children's Clinical University Hospital, Riga, Latvia
- Haukeland Universitetssykehus, Barneklinikken, Bergen, Norway
- Poland (2):
  - SPSK nr 1 im Prof. T Sokolowskiego, Szczecin
  - Instytut ''Pomnik - Centrum Zdrowia Dziecka'', Warsaw
- Russia (8):
  - Republic Children's Hospital of Ministry of Health of Udmurt, Izhevsk
  - Setchenov First Moscow State Medical University, Moscow
  - RMAPE, Moscow
  - Children's clinical city hospital #1, Novosibirsk
  - FSBEI of Higher Education "Rostov State Medical University", Rostov-on-Don
  - SPSBHI City Children out-patient clinic #44, Saint Petersburg
  - Samara Regional Children Clinical Hospital n.a. N.N. Ivanova, Samara
  - Siberian State Medical University, Tomsk
- Serbia (5):
  - University Children's Hospital Tirsova, Belgrade
  - Institute for Mother and Child Health Care of Serbia, Belgrade
  - University Clinical Centre Kragujevac, Kragujevac
  - Clinical Center in Nis, Niš
  - Institute for Health Care of Children and Adolescents, Novi Sad
- Spain (2):
  - Hospital Sant Joan de Déu, Esplugues Llobregat(Barcelona)
  - Hospital Clínico de Santiago de Compostela, Santiago de Compostela
- Switzerland (2):
  - Med. Kinder- und Poliklinik, Bern
  - Kinderspital Endokrinologie, Zürich, Zurich
- Thailand (3):
  - King Chulalongkorn Memorial hospital-Ped-Endocrinology, Bangkok
  - King Chulalongkorn Memorial hospital_Ped-Endocrinology, Bangkok
  - Phramongkutklao Hospital_Ped-Endo_Pediatrics, Bangkok
- Ukraine (3):
  - Dnipropetrovsk Regional Children's Clinical Hospital - Endocrinology department, Dnipro
  - Kharkiv Regional Children's Clinical Hospital - Endocrinological department, Kharkiv
  - Komisarenko Institute of Endocrinology and Metabolism of NAMSU - Department of paediatric endocrine pathology, Kyiv
- United Kingdom (4):
  - Hull Royal Infirmary_Hull, Hull
  - Alder Hey Children's Hospital, Liverpool
  - Royal London Hospital_London, London
  - Royal Manchester Children's Hospital, Manchester

IPD SHARING:
Plan to Share IPD: Yes
According to the Novo Nordisk disclosure commitment on novonordisk-trials.com
URL: http://novonordisk-trials.com

REFERENCES:
- [Derived] Juul A, Hojby M, Kawai M, Linglart A, Mori J, Zuckerman-Levin N, Backeljauw P. Somapacitan in children born small for gestational age: 4-year results from phase 2. Eur J Endocrinol. 2026 Feb 4;194(2):157-169. doi: 10.1093/ejendo/lvag017. PMID 41614610

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The trial was conducted at 38 sites in 12 countries as follows (number of sites that screened participants/ number of sites that randomized participants): Austria (2/1), France (2/2), Hungary (1/1), India (3/3), Israel (1/1), Italy (2/2), Japan (10/10), Latvia (1/1), Russia (6/6), Thailand (2/1), Ukraine (2/2) and United States (6/5).
Pre-assignment Details: Participants were randomized (1:1:1:1:1 ratio) to receive either once-weekly Somapacitan or daily Norditropin treatment during the main phase (26-week) and extension phase I (26-week). Followed by 208-week additional long-term safety extension phase (extension II) and a 30-day follow-up period. Results in this summary are reported based on main phase and extension phase I. The extension phase II is still ongoing and results will be posted after one year of study completion date.
Groups:
- Norditropin 0.035 mg/kg/Day: Participants received 0.035 mg/kg/day subcutaneous injection of norditropin daily during the main phase (26-week) and extension phase I (26-week).
- Norditropin 0.067 mg/kg/Day: Participants received 0.067 mg/kg/day subcutaneous injection of norditropin daily during the main phase (26-week) and extension phase I (26-week).
- Somapacitan 0.16 mg/kg/Week: Participants received 0.16 mg/kg/week subcutaneous injection of somapacitan once weekly during the main phase (26-week) and extension phase I (26-week).
- Somapacitan 0.20 mg/kg/Week: Participants received 0.20 mg/kg/week subcutaneous injection of somapacitan once weekly during the main phase (26-week) and extension phase I (26-week).
- Somapacitan 0.24 mg/kg/Week: Participants received 0.24 mg/kg/week subcutaneous injection of somapacitan once weekly during the main phase (26-week) and extension phase I (26-week).
Period: Overall Study
Arm/Group | Norditropin 0.035 mg/kg/Day | Norditropin 0.067 mg/kg/Day | Somapacitan 0.16 mg/kg/Week | Somapacitan 0.20 mg/kg/Week | Somapacitan 0.24 mg/kg/Week
Started | 12 | 13 | 12 | 13 | 12
Safety Analysis Set (SAS) (SAS included all randomized participants exposed to trial product.) | 12 | 13 | 12 | 13 | 12
Full Analysis Set (FAS) (FAS included all randomized participants exposed to the trial product.) | 12 | 13 | 12 | 13 | 12
Per Protocol Analysis Set (Participants from FAS who had not violated any inclusion/exclusion criteria and had used the randomized treatment for at least 22 weeks (for participants receiving Somapacitan) or 154 days (for participants receiving Norditropin).) | 11 | 13 | 12 | 13 | 12
Completed | 11 | 13 | 12 | 13 | 12
Not Completed | 1 | 0 | 0 | 0 | 0
Not completed — Withdrawn by parent or guardian | 1 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Full analysis set (FAS) included all randomized participants exposed to the trial product.
Groups:
- Total: Total of all reporting groups
Arm/Group | Norditropin 0.035 mg/kg/Day | Norditropin 0.067 mg/kg/Day | Somapacitan 0.16 mg/kg/Week | Somapacitan 0.20 mg/kg/Week | Somapacitan 0.24 mg/kg/Week | Total
Number analyzed (Participants) | 12 | 13 | 12 | 13 | 12 | 62
Age, Continuous [Mean (Standard Deviation); unit: years] | 6.29 (2.84) | 5.92 (2.44) | 6.13 (2.41) | 6.17 (2.21) | 6.00 (2.46) | 6.10 (2.39)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 4 | 4 | 4 | 4 | 22
  Male | 6 | 9 | 8 | 9 | 8 | 40
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 2 | 0 | 0 | 0 | 2
  Not Hispanic or Latino | 12 | 11 | 8 | 12 | 11 | 54
  Unknown or Not Reported | 0 | 0 | 4 | 1 | 1 | 6
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 9 | 8 | 4 | 7 | 6 | 34
  Asian | 3 | 5 | 6 | 4 | 6 | 24
  Other | 0 | 0 | 0 | 1 | 0 | 1
  Not reported | 0 | 0 | 2 | 1 | 0 | 3

OUTCOME MEASURES:

1. Primary Outcome: Height Velocity
Description: Height velocity (HV) was derived from height measurements taken at baseline (week 0) and week 26 visit as: HV = (height at 26 weeks visit - height at baseline)/(time from baseline to 26 weeks visit in years). The outcome measure was evaluated based on the data from in-trial observation period. In-trial observation period: from first administration and up until week 26 or last trial contact, whichever came first.
Time Frame: Baseline (week 0); week 26
Population: Full analysis set (FAS) included all randomized participants exposed to the trial product.
Measure: Mean (Standard Deviation); unit: centimeter per year (cm/year)
Arm/Group | Norditropin 0.035 mg/kg/Day | Norditropin 0.067 mg/kg/Day | Somapacitan 0.16 mg/kg/Week | Somapacitan 0.20 mg/kg/Week | Somapacitan 0.24 mg/kg/Week
Number analyzed (Participants) | 12 | 13 | 12 | 13 | 12
centimeter per year (cm/year) | 10.5 (2.0) | 11.9 (2.4) | 8.9 (1.8) | 11.1 (2.6) | 11.2 (3.4)
Statistical Analysis 1: Comparison: Norditropin 0.035 mg/kg/Day vs Somapacitan 0.16 mg/kg/Week; Test type: Superiority; Treatment difference = -1.4, 95% CI 2-sided [-3.2 to 0.4]
Statistical Analysis 2: Comparison: Norditropin 0.035 mg/kg/Day vs Somapacitan 0.20 mg/kg/Week; Test type: Superiority; Treatment difference = 0.7, 95% CI 2-sided [-1.1 to 2.5]
Statistical Analysis 3: Comparison: Norditropin 0.067 mg/kg/Day vs Somapacitan 0.20 mg/kg/Week; Test type: Superiority; Treatment difference = -0.9, 95% CI 2-sided [-2.6 to 0.9]
Statistical Analysis 4: Comparison: Norditropin 0.067 mg/kg/Day vs Somapacitan 0.24 mg/kg/Week; Test type: Superiority; Treatment difference = -0.6, 95% CI 2-sided [-2.4 to 1.2]

2. Secondary Outcome: Change in Ratio of Bone Age Versus Chronological Age
Description: Change in ratio of bone age (years) versus chronological age (years) from baseline (week 0) to week 52 is presented. X-rays of left hand and wrist for bone age assessment according to the Greulich and Pyle atlas were taken. X-ray images were sent to a central imaging laboratory for evaluation. Chronological Age (years) was calculated as: (Date minus Date of Birth) divided by 365.25. The outcome measure was evaluated based on the data from in-trial observation period. In-trial observation period: from first administration and up until week 52 or last trial contact, whichever came first.
Time Frame: Baseline (week 0); week 52
Population: Safety anslyis set (SAS) included all randomized participants exposed to the trial product. Overall number of participants analyzed = participants with available data for this outcome measure.
Measure: Mean (Standard Deviation); unit: ratio (bone age/chronological age)
Arm/Group | Norditropin 0.035 mg/kg/Day | Norditropin 0.067 mg/kg/Day | Somapacitan 0.16 mg/kg/Week | Somapacitan 0.20 mg/kg/Week | Somapacitan 0.24 mg/kg/Week
Number analyzed (Participants) | 11 | 13 | 12 | 11 | 12
ratio (bone age/chronological age) | -0.02 (0.13) | 0.07 (0.16) | 0.07 (0.08) | 0.03 (0.12) | -0.00 (0.10)

3. Secondary Outcome: Change in Height Standard Deviation Score (HSDS)
Description: Change in HSDS from baseline (week 0) to week 26 is presented. HSDS was derived using Centre for Disease Control and Prevention (CDC) standards. HSDS = [(height/population median)^skewness - 1]/(skewness * population standard deviation) where skewness, median and standard deviation is given by a reference growth table for the corresponding chronological age. The range for HSDS was -10 to +10. Negative scores indicated a height below the mean height for a child with the same age and gender, whereas positive scores indicated a height above the mean height for a child with the same age and gender. Positive value in change from baseline in HSDS indicated that HSDS was better than baseline HSDS In-trial observation period: from first administration and up until week 26 or last trial contact, whichever came first.
Time Frame: Baseline (week 0); week 26
Population: FAS included all randomized participants exposed to the trial product.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Norditropin 0.035 mg/kg/Day | Norditropin 0.067 mg/kg/Day | Somapacitan 0.16 mg/kg/Week | Somapacitan 0.20 mg/kg/Week | Somapacitan 0.24 mg/kg/Week
Number analyzed (Participants) | 12 | 13 | 12 | 13 | 12
score on a scale | 0.61 (0.19) | 0.73 (0.30) | 0.41 (0.20) | 0.66 (0.29) | 0.66 (0.37)

4. Secondary Outcome: Change in Height Velocity Standard Deviation Score (HVSDS)
Description: Change in HVSDS from baseline (week 0) to week 26 is presented. HVSDS was derived using Prader standards. HV SDS was calculated using the formula: HV SDS = (height velocity - mean)/standard deviation (SD), where height velocity was the height velocity variable measured, mean and SD of height velocity by gender and age for the reference population. The range for HVSDS was -10 to +10. Negative scores indicated a height velocity below the mean height velocity for a child with the same age and gender, whereas positive scores indicated a height velocity above the mean height velocity for a child with the same age and gender. Positive value in change from baseline in HVSDS indicated that HVSDS was better than baseline HVSDS. The outcome measure was evaluated based on the data from in-trial observation period. In-trial observation period: from first administration and up until week 26 or last trial contact, whichever came first.
Time Frame: Baseline (week 0); week 26
Population: FAS included all randomized participants exposed to the trial product.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Norditropin 0.035 mg/kg/Day | Norditropin 0.067 mg/kg/Day | Somapacitan 0.16 mg/kg/Week | Somapacitan 0.20 mg/kg/Week | Somapacitan 0.24 mg/kg/Week
Number analyzed (Participants) | 12 | 13 | 12 | 13 | 12
score on a scale | 6.37 (3.05) | 7.86 (1.88) | 4.03 (2.68) | 6.77 (3.35) | 7.24 (3.80)

5. Secondary Outcome: Change in Fasting Plasma Glucose
Description: Change in fasting plasma glucose from baseline (week 0) to week 26 is presented. The outcome measure was evaluated based on the data from on-treatment observation period. On-treatment observation period: from first administration and up until last trial contact, week 26 or 14 days after last administration, whichever came first.
Time Frame: Baseline (week 0); week 26
Population: Safety analysis set (SAS) included all randomized participants exposed to trial product.
Measure: Mean (Standard Deviation); unit: millimoles per liter (mmol/L)
Arm/Group | Norditropin 0.035 mg/kg/Day | Norditropin 0.067 mg/kg/Day | Somapacitan 0.16 mg/kg/Week | Somapacitan 0.20 mg/kg/Week | Somapacitan 0.24 mg/kg/Week
Number analyzed (Participants) | 12 | 13 | 12 | 13 | 12
millimoles per liter (mmol/L) | 0.382 (0.500) | 0.192 (0.415) | 0.167 (0.485) | 0.200 (0.912) | 0.275 (0.693)

6. Secondary Outcome: Change in Homeostatic Model Assessment for Steady State Beta Cell Function (HOMA-B)
Description: Change in HOMA-B from baseline (week 0) to week 26 is presented. HOMA-B is a measure of the beta cell function and was calculated as follows: HOMA-B = (20 * fasting insulin (picomoles per liter [pmol/L]) * 1/6(microunit per milliliter [µU/mL]))/ FPG(mmol/L)-3.5). HOMA-beta score ranges from minus infinity to infinity (no limits). Higher score means better beta-cell function for HOMA-beta. Negative change from baseline (week 0) in HOMA-B indicated a worse outcome. The outcome measure was evaluated based on the data from on-treatment observation period. On-treatment observation period: from first administration and up until last trial contact, week 26 or 14 days after last administration, whichever came first.
Time Frame: Baseline (week 0); week 26
Population: SAS included all randomized participants exposed to trial product. Overall number of participants analyzed = participants with available data for this outcome measure.
Measure: Mean (Standard Deviation); unit: HOMA-B index
Arm/Group | Norditropin 0.035 mg/kg/Day | Norditropin 0.067 mg/kg/Day | Somapacitan 0.16 mg/kg/Week | Somapacitan 0.20 mg/kg/Week | Somapacitan 0.24 mg/kg/Week
Number analyzed (Participants) | 12 | 13 | 12 | 13 | 11
HOMA-B index | 6.12 (99.55) | 63.35 (46.01) | 24.53 (49.59) | 0.75 (65.08) | 51.83 (88.89)

7. Secondary Outcome: Change in Homeostatic Model Assessment for Insulin Resistance (HOMA-IR)
Description: Change in HOMA-IR from baseline (week 0) to week 26 is presented. Insulin resistance is a condition in which cells fail to respond to normal actions of hormone in body. HOMA-IR is calculated using a participant's fasting plasma insulin and glucose levels. HOMA-IR = fasting serum insulin (micro international units per milliliter (μU/ml)) × fasting plasma glucose (millimoles per liter (mmol/l)) / 22.5. HOMA-IR scores are classified as follows: less than 1.0: considered insulin sensitive, 0.5-1.4: considered healthy, above 1.8: considered early insulin resistance; above 2.7 is considered significant insulin resistance. HOMA-IR score ranges from 0-infinity (no upper limit). Higher the score, higher the level of insulin resistance. The outcome measure was evaluated based on the data from on-treatment observation period. On-treatment observation period: from first administration and up until last trial contact, week 26 or 14 days after last administration, whichever came first.
Time Frame: Baseline (week 0); week 26
Population: SAS included all randomized participants exposed to trial product.
Measure: Mean (Standard Deviation); unit: HOMA-IR index
Arm/Group | Norditropin 0.035 mg/kg/Day | Norditropin 0.067 mg/kg/Day | Somapacitan 0.16 mg/kg/Week | Somapacitan 0.20 mg/kg/Week | Somapacitan 0.24 mg/kg/Week
Number analyzed (Participants) | 12 | 13 | 12 | 13 | 12
HOMA-IR index | 0.85 (0.82) | 1.17 (0.88) | 0.40 (0.48) | 0.57 (3.07) | 1.50 (2.10)

8. Secondary Outcome: Change in Glycated Haemoglobin (HbA1c)
Description: Change in HbA1c from baseline (week 0) to week 26 is presented. The outcome measure was evaluated based on the data from on-treatment observation period. On-treatment observation period: from first administration and up until last trial contact, week 26 or 14 days after last administration, whichever came first.
Time Frame: Baseline (week 0); week 26
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: Percentage of HbA1c
Arm/Group | Norditropin 0.035 mg/kg/Day | Norditropin 0.067 mg/kg/Day | Somapacitan 0.16 mg/kg/Week | Somapacitan 0.20 mg/kg/Week | Somapacitan 0.24 mg/kg/Week
Number analyzed (Participants) | 11 | 13 | 12 | 13 | 12
Percentage of HbA1c | -0.10 (0.39) | 0.03 (0.20) | 0.07 (0.15) | 0.12 (0.25) | 0.05 (0.24)

9. Secondary Outcome: Change in Insulin-like Growth Factor I (IGF-I) Standard Deviation Score (SDS)
Description: Change in IGF-I SDS from baseline (week 0) to week 26 is presented. IGF-I SDS was provided by the central laboratory; its calculation is based on the actual value of IGF-1 minus mean reference value of IGF-1 divided by reference standard deviation of IGF-1. The range for IGF-I SDS was from -10 to +10. Negative scores indicated a IGF-I below the mean IGF-I for a child with the same age and gender, whereas positive scores indicated a IGF-I above the mean IGF-I for a child with the same age and gender. Positive value in change from baseline in IGF-I SDS indicated that IGF-I SDS was higher than baseline IGF-I SDS. The outcome measure was evaluated based on the data from on-treatment observation period. On-treatment observation period: from first administration and up until last trial contact, week 26 or 14 days after last administration, whichever came first.
Time Frame: Baseline (week 0); week 26
Population: FAS included all randomized participants exposed to the trial product.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Norditropin 0.035 mg/kg/Day | Norditropin 0.067 mg/kg/Day | Somapacitan 0.16 mg/kg/Week | Somapacitan 0.20 mg/kg/Week | Somapacitan 0.24 mg/kg/Week
Number analyzed (Participants) | 12 | 13 | 12 | 13 | 12
score on a scale | 1.59 (0.67) | 2.13 (1.07) | 1.48 (0.90) | 1.93 (1.07) | 3.03 (1.42)

10. Secondary Outcome: Change in Insulin-like Growth Factor Binding Protein 3 (IGFBP-3) SDS
Description: Change in IGFBP-3 SDS from baseline (week 0) to week 26 is presented. The range for IGFBP-3 SDS was from -10 to +10. Negative scores indicated a IGFBP-3 below the mean IGFBP-3 for a child with the same age and gender, whereas positive scores indicated a IGFBP-3 above the mean IGFBP-3 for a child with the same age and gender. Positive value in change from baseline in IGFBP-3 SDS indicated that IGFBP-3 SDS was higher than baseline IGFBP-3 SDS. The outcome measure was evaluated based on the data from on-treatment observation period. On-treatment observation period: from first administration and up until last trial contact, week 26 or 14 days after last administration, whichever came first.
Time Frame: Baseline (week 0); week 26
Population: FAS included all randomized participants exposed to the trial product.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Norditropin 0.035 mg/kg/Day | Norditropin 0.067 mg/kg/Day | Somapacitan 0.16 mg/kg/Week | Somapacitan 0.20 mg/kg/Week | Somapacitan 0.24 mg/kg/Week
Number analyzed (Participants) | 12 | 13 | 12 | 13 | 12
score on a scale | 0.81 (0.64) | 1.06 (0.66) | 0.77 (0.68) | 1.01 (0.80) | 1.40 (0.88)

ADVERSE EVENTS:
Time Frame: From Baseline (Week 0) to Week 52
Description: All presented adverse events are treatment emergent adverse events (TEAEs) defined as an event that had onset after the first administration of trial product and up until 14 days after last trial drug administration for withdrawn participants, and with an onset after the first administration of trial product and up week 52. Results are based on the SAS which included all randomized participants exposed to trial product.
Groups:
- Norditropin (0.035mg/kg/Day): Participants received 0.035 mg/kg/day subcutaneous injection of norditropin daily during the main phase (26-week) and extension phase I (26-week).
- Norditropin (0.067mg/kg/Day): Participants received 0.067 mg/kg/day subcutaneous injection of norditropin daily during the main phase (26-week) and extension phase I (26-week).
- Somapacitan (0.16mg/kg/Week): Participants received 0.16 mg/kg/week subcutaneous injection of somapacitan once weekly during the main phase (26-week) and extension phase I (26-week).
- Somapacitan (0.20mg/kg/Week): Participants received 0.20 mg/kg/week subcutaneous injection of somapacitan once weekly during the main phase (26-week) and extension phase I (26-week).
- Somapacitan (0.24mg/kg/Week): Participants received 0.24 mg/kg/week subcutaneous injection of somapacitan once weekly during the main phase (26-week) and extension phase I (26-week).
Arm/Group | Norditropin (0.035mg/kg/Day) | Norditropin (0.067mg/kg/Day) | Somapacitan (0.16mg/kg/Week) | Somapacitan (0.20mg/kg/Week) | Somapacitan (0.24mg/kg/Week)
All-Cause Mortality (participants affected / at risk) | 0/12 | 0/13 | 0/12 | 0/13 | 0/12
Serious Adverse Events (participants affected / at risk) | 1/12 | 0/13 | 0/12 | 1/13 | 0/12
Other Adverse Events (participants affected / at risk) | 7/12 | 6/13 | 7/12 | 9/13 | 8/12
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Norditropin (0.035mg/kg/Day) (N=12) | Norditropin (0.067mg/kg/Day) (N=13) | Somapacitan (0.16mg/kg/Week) (N=12) | Somapacitan (0.20mg/kg/Week) (N=13) | Somapacitan (0.24mg/kg/Week) (N=12)
Inguinal hernia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Type 1 diabetes mellitus (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Norditropin (0.035mg/kg/Day) (N=12) | Norditropin (0.067mg/kg/Day) (N=13) | Somapacitan (0.16mg/kg/Week) (N=12) | Somapacitan (0.20mg/kg/Week) (N=13) | Somapacitan (0.24mg/kg/Week) (N=12)
Abdominal distension (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Anxiety (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Behaviour disorder (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bronchitis (Infections and infestations) | 0 (0) | 1 (3) | 0 (0) | 2 (4) | 0 (0)
Conjunctivitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 1 (3) | 0 (0) | 0 (0)
Dental caries (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Ear infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (2) | 1 (2) | 0 (0)
Enuresis (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 1 (1) | 1 (3) | 1 (1) | 0 (0)
Hypercholesterolaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hyperkalaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hyperkeratosis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Impaired fasting glucose (Metabolism and nutrition disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Influenza (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Influenza like illness (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Iron deficiency anaemia (Blood and lymphatic system disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nasopharyngitis (Infections and infestations) | 1 (1) | 1 (1) | 3 (6) | 2 (4) | 3 (5)
Otitis externa (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Otitis media (Infections and infestations) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Perioral dermatitis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pharyngitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Protein urine present (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 1 (1) | 0 (0) | 1 (4) | 1 (1) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Respiratory disorder (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (2) | 0 (0) | 1 (1) | 0 (0)
Respiratory tract infection viral (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Rhinitis (Infections and infestations) | 0 (0) | 1 (1) | 2 (6) | 0 (0) | 0 (0)
Stomatitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 2 (4) | 0 (0) | 2 (3) | 0 (0)
Varicella (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Viral infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 1 (3)
Vulvovaginal pruritus (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Allergy to arthropod bite (Immune system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Amblyopia (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Astigmatism (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Butterfly rash (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Contusion (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2)
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Eczema (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Erythema (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gastroenteritis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Growing pains (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hand dermatitis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Lipoatrophy (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Lymphadenitis (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Oral herpes (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Otitis media acute (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pallor (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Radius fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Respiratory syncytial virus infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Skin papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Urticaria (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
At the end of the trial, one or more scientific publications may be prepared collaboratively by the investigator(s) and Novo Nordisk. Novo Nordisk reserves the right to postpone publication and/or communication for up to 60 days to protect intellectual property.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-06-12): https://cdn.clinicaltrials.gov/large-docs/46/NCT03878446/Prot_SAP_000.pdf